CLINICAL TRIAL: NCT07200193
Title: A Multi-Center, Phase 1/2, Open-Label, Single and Multiple Ascending Dose Study of CRMA-1001 to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy in Adults With Chronic Hepatitis B
Brief Title: A Phase 1/2, Open-Label, Single and Multiple Ascending Dose Study of CRMA-1001 in Adults With Chronic Hepatitis B
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: nChroma Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRMA-1001-101
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepaititis B
Keywords: CHB; Chronic hepatitis B; Chronic HBV; Chronic Hep B; Chronic hepatitis; HBV
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CRMA-1001 Part A, SAD (Experimental): Single ascending dose arm
  Interventions: Genetic: CRMA-1001
- CRMA-1001 Part A, MAD (Experimental): Multiple ascending dose arm
  Interventions: Genetic: CRMA-1001
- CRMA-1001 Part B (Experimental): Dose expansion
  Interventions: Genetic: CRMA-1001

INTERVENTIONS:
Genetic: CRMA-1001 — Epigenetic gene silencing therapy delivered by intravenous (IV) infusion

SUMMARY:
This is an open-label study with single- and multiple-ascending dose arms followed by a dose expansion arm. The primary objective of the study is to determine the safety and tolerability of CRMA-1001 in adult participants with Chronic Hepatitis B. In addition, the pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of CRMA-1001 will be evaluated. CRMA-1001 is an epigenetic gene therapy delivered via intravenous (IV) infusion. Up to four dose levels will be tested. Participants will receive a single or multiple doses of CRMA-1001 and will remain on antiviral therapy during the dosing process.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female, weight 45-150 kg, age 18-64, inclusive
* Diagnosed with Chronic Hepatitis B
* On oral antiviral therapy
* ALT and AST <= 1.5 x ULN
* Total bilirubin <= ULN

Exclusion Criteria:

* Significant hepatic fibrosis or cirrhosis
* Current or prior liver disease other than HBV
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of CRMA-1001 | 6 months
  Incidence and severity of treatment-emergent adverse events

SECONDARY OUTCOMES:
Long-term safety of single and multiple doses of CRMA-1001 | 60 Months
  Incidence and severity of treatment emergent adverse events
Pharmacokinetics of CRMA-1001 components (Cmax) | 6 Months
  Maximum concentration (Cmax) in plasma
Pharmacokinetics of CRMA-1001 components (Tmax) | 6 Months
  Time of maximum concentration (Tmax) in plasma
Pharmacokinetics of CRMA-1001 components (terminal clearance rate) | 6 Months
  Clearance rate in terminal clearance phase (CL) in plasma
Pharmacokinetics of CRMA-1001 components (Vd) | 6 Months
  Volume of distribution (Vd) in plasma
To evaluate the immunogenicity of CRMA-1001 | 6 Months
  Incidence and characterization of anti-drug antibodies
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (HBsAg) | 6 Months
  Change from baseline in HBsAg
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (anti-HBs) | 6 Months
  Change from baseline in anti-HBs antibody titier
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (HBV DNA) | 6 Months
  Change from baseline in HBV DNA
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (HBeAg) | 6 Months
  Change from baseline in HBeAg
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (anti-HBe) | 6 Months
  Change from baseline in anti-HBe antibody titer
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (HBsAg) | 60 Months
  Change from baseline in HBsAg
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (anti-HBs) | 60 Months
  Change from baseline in anti-HBs antibody titer
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (HBV DNA) | 60 Months
  Change from baseline in HBV DNA
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (HBeAg) | 60 Months
  Change from baseline in HBeAg
To evaluate the effect of CRMA-1001 on circulating HBV biomarkers (anti-HBe) | 60 Months
  Change from baseline in anti-HBe antibody titer
To evaluate the rate of antiviral therapy discontinuation after treatment with CRMA-1001 | 60 Months
  Proportion of participants able to discontinue antiviral therapy
To evaluate the effect of CRMA-1001 on the incidence of functional cure | 60 Months
  Incidence of functional cure

CONTACTS AND LOCATIONS:
Locations (2):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No